CLINICAL TRIAL: NCT01442311
Title: Directly Observed Hepatitis C Treatment in Methadone Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-224; K23DA022454-01A1 (NIH)
Record Dates: First submitted 2011-09-27; First posted 2011-09-28 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C; Medication Adherence
Keywords: Hepatitis C Virus; Chronic Hepatitis C; Methadone; Injection Drug User; Adherence; Directly Observed Treatment
MeSH Terms: conditions — Hepatitis C; Medication Adherence; Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- enhanced DOT (PEG/RBV-DOT) (Experimental): Subjects randomized to the PEG/RBV-DOT arm receive weekly provider-administered pegylated interferon alfa-2a injections plus modified directly observed ribavirin therapy. We describe this as modified because ribavirin ingestion is observed at the methadone window three to six days per week based on the participants' methadone pick-up schedule, and only one of two daily doses is observed.
  Interventions: Other: enhanced DOT (both pegylated interferon alfa-2a and ribavirin)
- standard DOT (PEG-DOT) (Active Comparator): Subjects randomized to the Peg-DOT arm receive standard on-site treatment (weekly provider-administered pegylated interferon alfa-2a injections) and self-administered twice-daily oral ribavirin. Subjects in the PEG-DOT arm are dispensed monthly medication bottles of ribavirin, and ingest the ribavirin at home.
  Interventions: Other: standard DOT (PEG-DOT control arm)

INTERVENTIONS:
Other: enhanced DOT (both pegylated interferon alfa-2a and ribavirin) — Subjects randomized to the PEG/RBV-DOT arm receive weekly provider-administered pegylated interferon alfa-2a injections plus modified directly observed ribavirin therapy. We describe this as modified because ribavirin ingestion is observed at the methadone window three to six days per week based on the participants' methadone pick-up schedule, and only one of two daily doses is observed.
  Arms: enhanced DOT (PEG/RBV-DOT)
Other: standard DOT (PEG-DOT control arm) — Subjects randomized to the Peg-DOT arm receive standard on-site treatment (weekly provider-administered pegylated interferon alfa-2a injections) and self-administered twice-daily oral ribavirin. Subjects in the PEG-DOT arm are dispensed monthly medication bottles of ribavirin, and ingest the ribavirin at home.
  Arms: standard DOT (PEG-DOT)

SUMMARY:
Drug users account for a disproportionately large burden of hepatitis C virus (HCV) infection. However, HCV treatment adherence rates in drug users may be suboptimal in patients who use drugs regularly during HCV treatment. Because HCV treatment is most effective when patients adhere to at least 80% of the prescribed treatment regimen, interventions to improve HCV treatment adherence need to be developed and evaluated. The investigators designed the HCV DOT trial to test the efficacy of two versions of modified directly observed HCV therapy provided on-site at a methadone clinic. The primary objective of this trial is to determine whether enhanced DOT with both pegylated interferon alfa-2a plus ribavirin (PEG/RBV-DOT) is more efficacious than standard DOT with weekly provider-administered pegylated interferon (PEG-DOT) and self-administered ribavirin for increasing adherence and improving HCV treatment outcomes. The investigators hypothesize that PEG/RBV-DOT is associated with increased adherence and rates of sustained viral response compared with PEG-DOT.

ELIGIBILITY:
Inclusion Criteria:

* HCV-infected
* receive HCV medical care at the methadone clinic
* plan to initiate HCV treatment on-site within the next 3 months
* psychiatrically stable as determined by HCV treatment provider and/or on-site psychiatrist
* attend the methadone clinic between three and six days per week to receive methadone
* stable dose fo methadone for two weeks prior to the baseline visit

Exclusion Criteria:

* unable or unwilling to provide informed consent
* currently receiving HCV treatment
* primary HCV care provider does not agree to their participation in the trial
* psychiatrically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Adherence | 24 -48 weeks
  Adherence assessed by pill count, self-report, and medical records.

SECONDARY OUTCOMES:
sustained viral response (SVR) | 24 weeks after treatment completion
end of treatment response (ETR) | 24 - 48 weeks
treatment completion | 24 - 48 weeks
  completion of at least 80% of planned duration of HCV treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Litwin, MD, MPH, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine Division of Substance Abuse, The Bronx, New York, United States

REFERENCES:
- [Derived] Litwin AH, Berg KM, Li X, Hidalgo J, Arnsten JH. Rationale and design of a randomized controlled trial of directly observed hepatitis C treatment delivered in methadone clinics. BMC Infect Dis. 2011 Nov 12;11:315. doi: 10.1186/1471-2334-11-315. PMID 22078241